CLINICAL TRIAL: NCT06613997
Title: Randomized, Double-blind Trial Evaluating the Safety and Efficacy of a 21-day Course of Albendazole 400mg/Day in Subjects With High Loa Loa Microfilaremia
Brief Title: 21-day Double-blind Trial of Albendazole in Adults With Loa Loa Microfilaremia
Acronym: STOP-FiLAR-ALB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Programme National de Lutte contre l'Onchocercose, Republic of the Congo (Other Government)
Collaborators: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocole 129
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Loiasis With Positive Blood Microfilaremia; Loiasis
Keywords: filariasis; Albendazole; Onchocerciasis
MeSH Terms: conditions — Loiasis; Filariasis; Onchocerciasis | interventions — Albendazole

STUDY DESIGN:
Intervention Model Description: A 2-group, randomized, double-blind, parallel clinical trial:
  * albendazole 400 mg daily for 21 consecutive days
  * Placebo, daily for 21 consecutive days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albendazole 21 days (Experimental): Participants randomized in this arm will receive 21 days of albendazole 400mg/days .
  Interventions: Drug: Albendazole 400mg
- Placebo 21 days (Placebo Comparator): Participants randomized in this arm will receive 21 days of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole 400mg — Albendazole 400mg per days for 21 consecutive days
  Arms: Albendazole 21 days
Drug: Placebo — Placebo for 21 consecutive days
  Arms: Placebo 21 days

SUMMARY:
Our aim is to test the hypothesis that a 3-week course of albendazole 400 mg daily is safe and can progressively reduce Loa loa microfilarial densities in subjects with microfilaremia.

DETAILED DESCRIPTION:
Onchocerciasis, a parasitic disease caused by Onchocerca volvulus, present in sub-Saharan Africa, is subject of control programs based on the massive annual administration of ivermectin to the entire population living in endemic zones, without prior diagnosis. These programs are hampered in certain regions: areas coendemic with loasis (due to the Loa loa parasite) due to the risk of serious adverse effects caused by ivermectin in individuals heavily infected. The aim of this research is to evaluate an albendazole-based pre-treatment strategy to reduce the microfilarial density of loasis, enabling the safe use of ivermectin in all areas affected by onchocerciasis.

The efficacy of albendazole in reducing Loa loa microfilarial densities was evaluated in less than 100 individuals in 3 clinical trials. A 3-day regimen of ALB (200 mg daily) showed no effect on Loa loa microfilarial densities. A single dose of 800 mg every two months for one year induced a significant but insufficient reduction in Loa loa microfilarial densities to eliminate the risk of post-ivermectin side effects. The most interesting results came from a trial involving 21 subjects (10 in the albendazole group and 11 in the placebo group): twice-daily treatment with 200 mg ALB for 21 days progressively reduced Loa loa microfilarial densities by 80% over six months. However, the geometric mean of Loa loa microfilarial densities and the highest Loa loa microfilarial density in the albendazole group were 2,369 and 20,200 mf/mL respectively, i.e. below the risk threshold for serious adverse effects.

This project is based on a double-blind, randomized, placebo-controlled clinical trial. It aims to evaluate the safety and efficacy of 21 days of albendazole in Loa loa microfilaremia patients. The trial will be conducted in a rural area of Congo (Niari department, Mossendjo district and Lékoumou department, Komono district). A total of 100 subjects will be included in the study. Participants will receive either albendazole 400 mg daily or a similar placebo for 21 days. The aim is to recruit as many individuals as possible with at least 20,000 mfs/mL during the screening campaign, but we will be able to include all patients with microfilaremia. The individuals included will be monitored for 6 months (50 days of close follow-up for safety and 180 days of follow-up for efficacy). Initially, the majority of analyses will be descriptive. An Intention-to-Treat analysis will be performed. A Per Protocol analysis will be performed in the event of protocol deviations. The main evaluation criteria will be :

* Tolerance of a 21-day course of albendazole 400mg/day in L. loa-infected individuals with mfs in the bloodstream (criterion: no serious adverse events occurred in the albendazole-treated group).
* Efficacy: describe the kinetics of L. loa microfilarial densities (measured at 2, 7, 15, 22, 30, 90 and 180 days post-treatment) and the percentage of individuals who reduced their microfilarial load by at least 30% of their initial value.

The study will implement rigorous ethical procedures to ensure the safety and well-being of participants. The main objective is to minimize risks and maximize potential public health benefits. The study will comply with all applicable local laws, regulations and ethical guidelines (including the Declaration of Helsinki and Good Clinical Practice), and will be preceded by full information given to participants. Free and informed consent will be obtained, and participation will be voluntary. Risks include mild discomfort during the fingertip prick required for microfilaremia monitoring, and possible mild side effects associated with albendazole. On the other hand, benefits include the possibility of free medical screening and a contribution to medical research. Medical follow-up is planned to manage potential side effects. The research will be carried out in suitable, secure facilities, located close to the participating villages for assistance in the event of an emergency. A data anonymization system will be put in place to protect participants. Data will be secured on a server and exchanged securely. An Independent Monitoring Committee will oversee the study to guarantee the safety and interests of participants. Finally, specific insurance will cover participants in the event of study-related harm, ensuring adequate protection in the event of complications.

If successful, this project could revolutionize onchocerciasis control in areas coendemic with loasis. The proposed pre-treatment strategy could enable ivermectin to be administered safely, helping to speed up the elimination of onchocerciasis. In addition, this project could have important implications for the individual treatment of subjects with high Loa loa microfilarial density, offering an alternative to currently complicated and ineffective treatments.

ELIGIBILITY:
Inclusion Criteria:

* Consent informed, written, signed and dated
* Women or men aged 18 to 70 years inclusive
* Carrier of L. loa microfilaremia
* Body weight ≥ 40 kg and less than 90 kg

Exclusion Criteria:

* Participation in any study other than a purely observational study, within the 4 weeks preceding this study (determined by the theoretical date of the first administration of albendazole placebo)
* Any vaccination within 4 weeks previous to this study
* Infection requiring treatment in the 10 days previous to this study, as determined by the anamnesis during the medical interview (e.g. pulmonary infection , digestive or skin infection; with or without antibiotic treatment)
* Known immunosuppressive pathology (by self-report)
* Past or present history of neurological (including epilepsy) or neuropsychiatric disease
* Current treatment with ritonavir and/or rifampicin
* Use of cocaine or other drugs of abuse in the 72 hours preceding administration of the trial treatment, as determined by history during the medical interview
* Past or present history of liver, kidney or bone marrow failure
* ALAT transaminase level ≥ 3 times the upper limit of normal (3N) according to laboratory standards
* Any condition, in the opinion of the investigator, that exposes the subject to undue risk
* Known intolerance to ALB or benzimidazole derivatives in general
* Subjects who donated blood in the previous 8 weeks to study entry, with a standard volume (500 mL)
* On clinical examination: symptoms, physical signs or laboratory findings suggestive of systemic disorders, including disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other abnormalities that could interfere with the interpretation of trial results. The physician may then give a favorable or unfavorable opinion on the participants inclusion.
* ALB and/or mebendazole in the last month
* IVM taken in the last month
* Any condition which, in the opinion of the investigator, exposes the subject to undue risk
* Positive urine pregnancy test for women of childbearing age or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerance of Albendazole 400mg/day in individuals with Loa loa microfilaremia | During the treatment (21 days) and 3 month after
  The proportion of AEs and/or SAEs occurring in the treatment (ALB) and placebo groups and the proportion of AEs and/or SAEs occurring by grade in the treatment (ALB) and placebo groups
Efficacity of Albendazole 400mg/day in individuals with Loa loa microfilaremia | During the treatment (21 days) and 6 months after
  Rate of reduction of L. loa DMF in blood at D2, D7, D15, D22, D30, D90 and D180 in each of the two groups and proportion of subjects without L. loa microfilariae in blood at D2, D7, D15, D22, D30, D90 and D180 in both groups

SECONDARY OUTCOMES:
Comparison the safety of albendazole to placebo in individuals with Loa loa microfilaremia | From Day 2 after the first dose to 6 months after the first dose
  Comparison of occurrence of adverse events by proportion and grade in treatment group (ALB) and placebo group and comparison of DMF reduction rates in L. loa during treatment (D1 to D21) and those observed over the long term (D21 to D180)

CONTACTS AND LOCATIONS:
Overall Officials: Jéremy CAMPILLO, PharmD PhD, Study Director — Institut de Recherche pour le Développement (IRD); François MISSAMOU, MD, Principal Investigator — Programme National de Lutte contre l'Onchocercose (PNLO)

IPD SHARING:
Plan to Share IPD: No